CLINICAL TRIAL: NCT02188901
Title: Contrast (Sonazoid)-Enhanced US as a Screening Tool for Hepatocellular Carcinoma in Cirrhosis: An Exploratory Cross-sectional Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 4-2014-0337
Record Dates: First submitted 2014-07-03; First posted 2014-07-14 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: HCC; Sonazoid; Ultrasonography; Screening
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm (Other)
  Interventions: Other: Sonazoid-enhanced ultrasonography

INTERVENTIONS:
Other: Sonazoid-enhanced ultrasonography — Sonazoid (perflubutane) [GE healthcare]
  Other Names: 0.015ml/kg of suspension containing 16μl of perflubutane microbubble and 2ml of diluent, IV (in the vein) on day 1

SUMMARY:
B-mode ultrasonography (B-US), a standard method of surveillance of hepatocellular carcinoma (HCC), has a fair sensitivity of 63% in detecting early stage HCC. Sonazoid, a contrast agent for ultrasonography, has reported to have superior sensitivity in detecting focal liver lesion since it has ability of Kupffer phase imaging as well as vascular phase imaging. So our aim is to compare the detection rate of early stage HCC and false referral rate of HCC between B-mode US and Sonazoid-enhanced ultrasonography (S-US) within the same prospective data group. Our hypothesis is that S-US has superior detection rate of early stage HCC (5%) than that of B-mode US (3%).

ELIGIBILITY:
Inclusion Criteria:

1. Patient 20 years old or older,
2. Patient at high risk of HCC and is supposed to take ultrasonography,
3. Patient who has no suspicious HCC on previous examinations or patient who undergoes the first surveillance,
4. Patient who has liver cirrhosis proven by one of the following methods-liver biopsy (METAVIR score 4), identification of esophageal or gastric varix by endoscopically or radiologically, surface nodularity on ultrasonography, CT or MRI, platelet count less than 100,000/mm3, serum albumin less than 3.5 g/dl, or prothrombin time higher than 1.3 INR,
5. Patient without contraindication for sonazoid,
6. Patient willing to sign the informed consent

Exclusion Criteria:

1. Patient on pregnancy or breast feeding,
2. Patient with allergy to egg,
3. Patient with left-to-right shunt, respiratory insufficiency, or severe pulmonary hypertension,
4. Patient with history of HCC,
5. Patient with history of malignancy other than HCC -

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 523 (Actual)
Dates: Start 2014-10-15 (Actual); Primary Completion 2016-08-03 (Actual); Study Completion 2016-08-03 (Actual)

PRIMARY OUTCOMES:
Detection rate of early stage HCC | 30±30 days after S-US if there is one or more suspicious HCC detected on S-US, or 180±30 days after S-US if there is no suspicious HCC detected on S-US
  Detection rate of early-stage HCC = (Number of confirmed early-stage HCC detected by a given modality) / (Total number of patients enrolled) x100
False referral rate of HCC | 30±30 days after S-US if there is one or more suspicious HCC detected on S-US, or 180±30 days after S-US if there is no suspicious HCC detected on S-US
  False referral rate of HCC =

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Park JH, Park MS, Lee SJ, Jeong WK, Lee JY, Park MJ, Lee SS, Han K, Nam CM, Park SH, Lee KH. Contrast-enhanced US with Perfluorobutane for Hepatocellular Carcinoma Surveillance: A Multicenter Diagnostic Trial (SCAN). Radiology. 2019 Sep;292(3):638-646. doi: 10.1148/radiol.2019190183. Epub 2019 Jul 9. PMID 31287387
- [Derived] Park JH, Park MS, Lee SJ, Jeong WK, Lee JY, Park MJ, Han K, Nam CM, Park SH, Lee KH. Contrast-enhanced US with Perfluorobutane(Sonazoid) used as a surveillance test for Hepatocellular Carcinoma (HCC) in Cirrhosis (SCAN): an exploratory cross-sectional study for a diagnostic trial. BMC Cancer. 2017 Apr 18;17(1):279. doi: 10.1186/s12885-017-3267-8. PMID 28420329